CLINICAL TRIAL: NCT05679362
Title: How 2 Deal With PCOS: a Randomized Online Intervention for Women With PCOS
Brief Title: Online Brief CBT Intervention for Women With PCOS
Acronym: How2deal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: The Waterloo Foundation (Other)
Responsible Party: Principal Investigator, Geranne Jiskoot, Principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: How2deal
Record Dates: First submitted 2022-12-16; First posted 2023-01-11 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries; Depression, Anxiety; Self Esteem
MeSH Terms: conditions — Polycystic Ovary Syndrome; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- immediate individual treatment (A) (Experimental): 5 online individual sessions
  Interventions: Behavioral: online brief CBT intervention
- immediate group treatment (B) (Experimental): 5 online group sessions with other women with PCOS
  Interventions: Behavioral: online brief CBT intervention
- care as usual (cau) (No Intervention): The CAU group receives standard treatment for depressive symptoms from their general practitioner (GP).

INTERVENTIONS:
Behavioral: online brief CBT intervention — Cognitive behavioral therapy
  Arms: immediate group treatment (B); immediate individual treatment (A)

SUMMARY:
Primary Objective:

-To study if an online individual brief CBT (group A) intervention is effective for psychological distress (anxiety and depression) compared to a CAU group in patients with PCOS at 3 and 6 months relative to baseline.

Secondary Objective(s):

1. To study if an online group based brief CBT (group B) is more effective for anxiety and depression compared to CAU in patients with PCOS at 3 and 6 months relative to baseline.
2. To determine if an online individual brief CBT (group A) is effective for improvements in QoL, coping strategies, body image and sleep quality compared to CAU in patients with PCOS at 3 and 6 months relative to baseline.
3. To determine if an group based brief CBT (group B) is more effective for improvements in QoL, coping strategies, body image and sleep quality compared to CAU in patients with PCOS at 3 and 6 months relative to baseline.
4. If A and B are effective compared to CAU, we will compare online individual brief CBT (group A) to online group based brief CBT (group B) for anxiety and depression, QoL, coping strategies, body image and sleep quality compared to in patients with PCOS at 3 and 6 months relative to baseline.

DETAILED DESCRIPTION:
The online brief CBT intervention is designed to address three problems that have often been reported in women with PCOS. Therefore, the program contains three themes: Psychoeducation about PCOS; traditional CBT and problem-solving therapy.

Participants are randomized into one of three groups:

1. individual treatment (A)
2. group treatment (B)
3. care as usual (CAU)

Treatment A and B include 5 sessions divided over a period of 3 months:

Week 1: Session 1 +homework assignments Week 3: Session 2 +homework assignments Week 5: Session 3 +homework assignments Week 8: Session 4 +homework assignments Week 12: Session 5 +homework assignments

The CAU group receives standard treatment for depressive symptoms from their general practitioner (GP).

ELIGIBILITY:
Inclusion Criteria:

* women with a confirmed diagnosis of PCOS based on the Rotterdam criteria
* body Mass Index (BMI) ≥18.5 kg/m2
* aged 18-55 years.
* mild depressive symptoms or anxiety scores based on the Hospital Anxiety and Depression Scale (HADS) and/or a negative body image based on the Body Cathexis Scale (BCS).

Exclusion Criteria:

* pregnancy
* current treatment for clinical depression, anxiety disorders or eating disorders
* suicidality (indicated by a score >2 on the Beck Depression Inventory II suicide item)
* having an endocrine disease (diabetes mellitus, thyroid function disorders, Cushing's disease, adrenal tumors, and congenital adrenal hyperplasia)
* inability to speak, read or write Dutch.

Ages: 17 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Gender identity
Enrollment: 222 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Depression | at start, after 3 and 6 months
  Changes in depression scores as assessed by the Hospital anxiety and depression scale (HADS). HADS is a 14-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression. A higher score indicates higher distress.
Anxiety | at start, after 3 and 6 months
  Changes in anxiety scores as assessed by the Hospital anxiety and depression scale (HADS). HADS is a 14-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression. A higher score indicates higher distress.

SECONDARY OUTCOMES:
QoL | at start, after 3 and 6 months
  The Polycystic Ovary Syndrome Quality of Life scale (PCOSQOL). The PCOSQOL is a 35-item questionnaire with four subscales: Impact of PCOS, Infertility, Hirsutism and Mood. Lower scores represent a decreased QoL.
Coping | at start, after 3 and 6 months
  Coping Inventory for stressful situation (CISS). Scores for all items per scale are summed to form scale scores; higher scores indicate a greater use of that particular coping strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided